CLINICAL TRIAL: NCT03139253
Title: Antimicrobial Susceptibility Testing Guided Triple Therapy in Salvage Helicobacter Pylori Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Organization: Shandong University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017SDU-QILU-02
Record Dates: First submitted 2017-04-23; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Antimicrobial Susceptibility Testing; Triple Therapy
Keywords: Helicobacter Pylori Infection; Antimicrobial susceptibility testing (AST); Triple Therapy
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Tinidazole; Levofloxacin; Furazolidone; Tetracycline; ilaprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- clarithromycin susceptible (Experimental): Patients will receive a 14-day triple therapy to eradicate H. pylori. The regimen is consist of Ilaprazole, amoxicillin and clarithromycin.
  Ilaprazole 5 mg b.i.d is used as the proton pump inhibitor (PPI).
  Interventions: Drug: amoxicillin; Drug: clarithromycin; Drug: Ilaprazole
- metronidazole susceptible (Experimental): Patients will receive a 14-day triple therapy to eradicate H. pylori. The regimen is consist of Ilaprazole, amoxicillin and tinidazole.
  Interventions: Drug: amoxicillin; Drug: tinidazole; Drug: Ilaprazole
- levofloxacin susceptible (Experimental): Patients will receive a 14-day triple therapy to eradicate H. pylori. The regimen is consist of Ilaprazole, amoxicillin and levofloxacin.
  Interventions: Drug: amoxicillin; Drug: levofloxacin; Drug: Ilaprazole
- furazolidone susceptible (Experimental): Patients will receive a 14-day triple therapy to eradicate H. pylori. The regimen is consist of Ilaprazole, amoxicillin and furazolidone.
  Interventions: Drug: amoxicillin; Drug: furazolidone; Drug: Ilaprazole
- tetracycline susceptible (Experimental): Patients will receive a 14-day triple therapy to eradicate H. pylori. The regimen is consist of Ilaprazole, amoxicillin and tetracycline.
  Interventions: Drug: amoxicillin; Drug: tetracycline; Drug: Ilaprazole

INTERVENTIONS:
Drug: amoxicillin — amoxicillin 1000 mg bid. for 14 days
Drug: clarithromycin — clarithromycin 500 mg bid. for 14 days.
  Arms: clarithromycin susceptible
Drug: tinidazole — tinidazole 500 mg bid. for 14 days.
  Arms: metronidazole susceptible
Drug: levofloxacin — levofloxacin 500 mg qd. for 14 days.
  Arms: levofloxacin susceptible
Drug: furazolidone — furazolidone 100 mg bid. for 14 days.
  Arms: furazolidone susceptible
Drug: tetracycline — tetracycline 750 mg bid. for 14 days.
  Arms: tetracycline susceptible
Drug: Ilaprazole — Ilaprazole 5 mg bid. for 14 days.

SUMMARY:
Helicobacter pylori (H. pylori), which infects about 50% of the global population, has been recognized as a main risk factor of multiple gastric pathologies, especially non-cardiac gastric cancer. Strongly evidence supports that H. pylori eradication is an effective approach to reduce the incidence of those pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who are 18-70 years old with persistent H. pylori infection after first or second line treatment attempts.

Exclusion Criteria:

* Enable to undergo upper endoscopy;
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Known or suspected allergy to study medications;
* Taking bismuth and antibiotics in the previous four weeks, or taking proton pump inhibitor and H2-receptor blockers in the previous two weeks;
* Currently pregnant or lactating
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of AST guided triple therapy | 3 months

SECONDARY OUTCOMES:
the rate of improving dyspepsia symptoms after H. pylori eradication | 3 months
the rate of adverse events happening | 3 months
the rate of good compliance (take pills more than 90%) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No